CLINICAL TRIAL: NCT02180321
Title: Effect of Tranexamic Acid Based on Pharmacokinetics in Pediatric Patients Undergoing Craniosynostosis Surgery: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2014-0274
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Craniosynostosis Patients Undergoing Distraction Osteotomy
Keywords: Tranexamic acid; pharmacokinetics; craniosynostosis
MeSH Terms: conditions — Craniosynostoses | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Drug: normal saline
- Tranexamic acid (Experimental)
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — 10mg/kg of tranexamic acid loading infusion for 15 min from beginning of the surgery, then continuous infusion throughout the surgery for 5mg/kg/hr
  Arms: Tranexamic acid
Drug: normal saline — 10mg/kg of normal saline loading infusion for 15 min from beginning of the surgery, then continuous infusion throughout the surgery for 5mg/kg/hr
  Arms: Control

SUMMARY:
Massive bleeding is expected when performing distraction osteotomy for craniosynostosis patients. Since such operation is performed at very young age, many efforts are performed in order to reduce the total amount of bleeding and the transfusion during and after the surgery. Our study aims at correcting the coagulopathy from massive bleeding and transfusion during distraction osteotomy using continuous infusion of antifibrinolytic agent, tranexamic acid. Tranexamic acid infusion is determined according to the pharmacokinetic model, and the changes in coagulopathy will be defined using thromboelastography.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for distraction osteostomy under the diagnosis of Craniosynostosis.
2. Patients aged from 2 months to 6 years, either of whose patients had consented
3. ASA class 1 or 2

Exclusion Criteria:

1. Coagulopathy with either PT > INR 1.5 or PLT < 50,000/dL
2. Patients took any NSAIDs within 2 days, or aspirin within 14 days prior to surgery
3. History of convulsive seizure, epilepsy, any brain surgery
4. Known drug allergic reaction to tranexamic acid

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Bleeding loss | from every each hour during intraop, periodImmediate postop, postoperative 24hr to postoperative 48hr
  Assessing the amount of bleeding during each intraop hours, and postoperative periods.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University College of Medicine, Seoul, Seoul, South Korea